CLINICAL TRIAL: NCT05266287
Title: Evaluating Changes in Microbiota Composition and Quality of Life in Irritable Bowel Syndrome: A Randomized, Controlled Trial
Brief Title: Changes in Microbiota and Quality of Life in IBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Ryan Bradley, Director of Research, National University of Natural Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RB120721
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational supplement (Experimental): Participants in this arm will take a supplement containing 2'-fucosyllactose (2'-FL)
  Interventions: Dietary Supplement: a supplement containing 2'-fucosyllactose (2'-FL)
- Placebo supplement (Placebo Comparator): Participants in this arm will take a placebo supplement
  Interventions: Dietary Supplement: Placebo Supplement

INTERVENTIONS:
Dietary Supplement: a supplement containing 2'-fucosyllactose (2'-FL) — Participants will be asked to take a commercially available dietary supplement containing 833 mg of 2'-FL, 220 mg of a blend of organic beet root and okra fruit, 100 mg of Collinsonia root, 37.5 mg organic rice hull concentrate, and 14 mg calcium stearate.
  Arms: Investigational supplement
Dietary Supplement: Placebo Supplement — Participants will be asked to take a placebo supplement containing 510.9 mg organic sucanat, 385.4 mg calcium phosphate, 304.7 mg cellulose, 143.4 mg date powder, 39.4 mg rice bran powder, 9.0 mg gum arabic, and 7.2 mg calcium stearate.
  Arms: Placebo supplement

SUMMARY:
The primary research question to be addressed is: Does a 2'-FL-containing dietary supplement impact stool microbiota composition in adults with IBS? The primary measure for determining potential impacts of the 2'-FL-containing dietary supplement on stool microbiota composition is stool abundance of Faecalibacterium prausnitzii, a commensal intestinal bacteria. Additional measures related to determining potential impacts of the 2'-FL-containing dietary supplement on gut microbiota composition are stool levels of additional commensal intestinal bacteria and measures of intestinal microbial diversity.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-70 years (inclusive)
* Existing diagnosis of IBS
* Willing to take the 2'-FL-containing dietary supplement (or a control supplement) three times per day for 6 weeks
* Willing to attend 4 in-person study visits
* Willing to collect 3 stool samples at home
* Willing to periodically monitor stool form/consistency (and log the information on a diary)
* Willing to complete IBS symptom focused questionnaires
* Willing to refrain from making changes in dietary supplements and medications for the duration of the study
* Willing to maintain current dietary pattern for the duration of the study
* Willing to maintain current exercise pattern for the duration of the study
* Able to speak, read, and understand the English language
* Able to provide written informed consent

Exclusion Criteria:

* Do not have an active primary care provider or specialist managing their IBS
* Initiation of or changes to supplements or medications within 2 weeks prior to screening and/or enrollment (changes include stopping or changing the dose of supplements or medications)
* Intake of prebiotic or fiber supplement(s) (current intake or intake within 2 weeks prior to screening and/or enrollment)
* Intake of probiotic supplement(s) (current intake or intake within 2 weeks prior to screening and/or enrollment)
* Use of antibiotic, antiparasitic, or antifungal medications orally or intravenously (current use or use within 2 weeks prior to screening and/or enrollment)
* Initiation of or changes to an exercise regimen within 2 weeks prior to screening and/or enrollment
* Initiation of or changes to a food plan within 2 weeks prior to screening and/or enrollment
* Current involvement or within 2 weeks prior to screening and/or enrollment of a significant diet or weight loss program (such as NutriSystem, Jenny Craig, Atkin's or other low-carb diet programs) or very low-calorie liquid diet programs (such as Optifast, Medifast, and/or HMR)
* Current or previous history of chronic gastrointestinal illness other than IBS (e.g. inflammatory bowel disease, celiac disease, diverticulitis, cirrhosis, hepatitis, etc.)
* History of gastrointestinal surgery other than appendectomy (e.g. weight loss surgery, cholecystectomy, splenectomy, etc.)
* Major medical or surgical event requiring hospitalization (for any reason other than a minor scheduled medical procedure) within 3 months prior to screening
* Cancer diagnosis or treatment within the last 5 years (with the exception of basal cell carcinoma, squamous cell carcinoma, and/or carcinoma in situ of the cervix)
* Currently participating in another interventional research study or participated in another interventional study within 2 weeks prior to screening
* Known intolerance or allergy to ingredients that may be in the study supplement or control supplement (Collinsonia root, beet root, okra, date powder, sucanat, rice hull concentrate, rice bran extract, cellulose, calcium stearate, calcium phosphate, gum arabic, or a trace amount of lactose)
* Women who are lactating, pregnant or planning pregnancy within the next 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
F. Prausnitzii abundance | 6 weeks
  F. Prausnitzii abundance will be measured in stool via 16s RNA sequencing and quantified

SECONDARY OUTCOMES:
F. Prausnitzii relative abundance | 6 weeks
  F. Prausnitzii abundance will be measured in stool via 16s RNA sequencing and the proportion to other organisms calculated
Bifidobacterium spp. relative abundance | 6 weeks
  Bifidobacterium spp. relative abundance in stool will be measured via 16s RNA sequencing and the proportion to other organisms calculated
Alpha diversity of the microbiota | 6 weeks
  Alpha diversity is a measure of overall diversity of organisms within in a stool sample
Beta diversity of the microbiota | 6 weeks
  Beta diversity is a measure of overall diversity of organisms between stool samples in the cohort of participants
IBS-Severity Scoring System | 6 weeks
  Validated instrument that quantified patient-reported IBS severity
IBS-Adequate Relief from Symptoms | 6 weeks
  Validated instrument that measures patient-reported relief from IBS symptoms
Bristol Stool Form Scale | 6 weeks
  7-point scale used qualitatively assessing form of stool

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Bradley, ND, MPH, Principal Investigator — National University of Natural Medicine
Locations (1):
- National University of Natural Medicine, Portland, Oregon, United States